CLINICAL TRIAL: NCT03569670
Title: All-Polyethylene Tibial Components in Total Knee Arthroplasty: A Radiostereometric Analysis Comparing Posterior Stabilizing and Condylar Stabilizing Implants
Brief Title: All-Polyethylene Tibias in TKA: PS vs CS Implants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been suspended due to inability to obtain funding.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110812
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis, Knee
Keywords: cost; total knee replacement; arthroplasty; posterior stabilized; cruciate retaining; all-polyethylene
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Stabilized (Experimental): A posterior stabilized, all-polyethylene tibial component will be used during surgery.
  Interventions: Device: Posterior stabilized all-polyethylene tibial component
- Cruciate Retaining (Active Comparator): A cruciate retaining, all-polyethylene tibial component will be used during surgery.
  Interventions: Device: Cruciate retaining all-polyethylene tibial component

INTERVENTIONS:
Device: Posterior stabilized all-polyethylene tibial component — Patients randomized to this arm will have a Triathlon implant with a posterior stabilized, all-polyethylene tibial component used during surgery.
  Arms: Posterior Stabilized
Device: Cruciate retaining all-polyethylene tibial component — Patients randomized to this arm will have a Triathlon implant with a cruciate retaining, all-polyethylene tibial component used during surgery.
  Arms: Cruciate Retaining

SUMMARY:
This is a randomized control trial where patients will be randomized to receive one of two types of total knee arthroplasty (TKA) all-polyethylene (AP) tibial components: cruciate retaining (CR) or posterior stabilized (PS). We will use radiostereometric analysis to assess the stability of the implants at 6 weeks, 3 months, 6 months, 1 year and 2 year post-operatively. The main objective of this project will be to determine which AP tibial component offers the greatest stability. Additionally, we will seek to determine whether patient BMI significantly impacts the stability of AP tibial components.

DETAILED DESCRIPTION:
With healthcare expenditures rising as our population ages, there have been significant efforts targeted towards streamlining costs associated with various medical treatments. One area of substantial spending in the orthopaedic surgery field is total joint replacements. The effort to reduce costs has sparked a renewed interest in the use of allpolyethylene (AP) tibial components in total knee arthroplasty (TKA).

In recent years, there has been ample research demonstrating that AP tibial components have performed as good as, or better, than metal-backed (MB) tibial components. Some studies have estimated that cost savings could be as high as 50% with routine use of AP tibial components. While sufficient literature exists demonstrating the equivalence or superiority of AP versus MB designs, there is a paucity of work done comparing different types of AP tibial components.

Tibial components in TKA can be of the posterior stabilizing (PS) or cruciate retaining (CR) variety. To date, we are unaware of any study that directly compares AP tibial PS components to AP tibial CR components.

Radiostereometric analysis (RSA) has evolved as an exceptionally precise and reliable method for assessing the migration of components in total joint arthroplasty. Using RSA data, it is possible to accurately predict, within the first 24 months post-operatively, the survival of a total joint arthroplasty. Furthermore, the use of RSA outcomes in arthroplasty research allows for adequately powered studies with significantly smaller sample sizes than previously required.

The main objective of this project will be to determine which AP tibial component offers the greatest stability. Additionally, we will seek to determine whether patient body mass index (BMI) significantly impacts the stability of AP tibial components.

We will prospectively enroll patients who will be undergoing a total knee arthroplasty by one of the study investigators. Potentially eligible patients will have the project explained to them during their preadmission clinic visit prior to surgery and if interested a member of the research team will perform the informed consent process. Should a patient elect to participate in the study they will sign the informed consent form and complete demographics and baseline health related quality of life questionnaires including Oxford Knee, EQ-5D, and the VR-12, in addition to the Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) which is already completed as per standard of care. The baseline demographic characteristics that will be collected include age, BMI, gender, and relevant medical comorbidities. Patients will be randomized to have either a PS or CR all-poly tibial component used during surgery. Randomization will be stratified by BMI to ensure equal distribution in both groups.

During surgery the surgeon will insert 6-9 tantalum beads in the proximal tibial, 6 beads in the polyeythylene tray, and another bead into the tip of the polyethylene stem. These beads will be used to measure migration of the implants on RSA imaging (radiostereometric analysis).

The RSA x-rays will be taken at baseline (2 weeks) and at the 6-week, 3 months, 6 months and 1 year and 2 year follow-up appointments. These images will be taken at Robarts Research Institute in the RSA analysis suite. At the 3month, 6 month, 1 year and 2 year visits we will also collect health related quality of life questionnaires including the WOMAC, Oxford Knee, EQ-5D and the VR-12.

Patients and data collector will be blinded to treatment arm. The person who will analyze the RSA images will be able to see which treatment arm participants belong to (based on viewing xrays) however the hypothesis of the study will not be revealed to them prior to analysis.

Intra-operative cost information will also be collected using institutional cost data in order to compare differences in OR costs between the two implant designs and across BMI categories.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis
* primary total knee arthroplasty
* able to consent for themself

Exclusion Criteria:

* inflammatory arthropathy
* fibromyalgia
* chronic pain syndrome
* previous distal femur or proximal tibia open reduction internal fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Implant Migration | Change between baseline (taken at 2 weeks post-operatively) and 2 years
  Comparison of the two component types using radiostereometric analysis imaging.

SECONDARY OUTCOMES:
VR-12 | 2 years
  Patient-reported outcome used to assess general health.
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | 2 years
  Patient-reported outcome used to assess function, pain and stiffness.
Oxford Knee Score | 2 years
  Patient-reported outcome used to assess knee function.
EQ-5D | 2 years
  Patient-reported outcome used to assess quality of life.
Cost | Intraoperative
  Intraoperative costs will be collected using institutional cost data.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Vasarhelyi, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Gioe TJ, Maheshwari AV. The all-polyethylene tibial component in primary total knee arthroplasty. J Bone Joint Surg Am. 2010 Feb;92(2):478-87. doi: 10.2106/JBJS.I.00842. PMID 20124081
- [Background] Medel F, Kurtz SM, Klein G, Levine H, Sharkey P, Austin M, Kraay M, Rimnac CM. Clinical, surface damage and oxidative performance of poly II tibial inserts after long-term implantation. J Long Term Eff Med Implants. 2008;18(2):151-65. doi: 10.1615/jlongtermeffmedimplants.v18.i2.40. PMID 19968624
- [Background] Adalberth G, Nilsson KG, Bystrom S, Kolstad K, Milbrink J. Low-conforming all-polyethylene tibial component not inferior to metal-backed component in cemented total knee arthroplasty: prospective, randomized radiostereometric analysis study of the AGC total knee prosthesis. J Arthroplasty. 2000 Sep;15(6):783-92. doi: 10.1054/arth.2000.8101. PMID 11021456
- [Background] Yassin M, Garti A, Weissbrot M, Ashkenazi U, Khatib M, Robinson D. All-polyethylene tibial components are not inferior to metal-backed tibial components in long-term follow-up of knee arthroplasties. Eur J Orthop Surg Traumatol. 2015 Aug;25(6):1087-91. doi: 10.1007/s00590-015-1645-y. Epub 2015 May 26. PMID 26006786
- [Background] Norgren B, Dalen T, Nilsson KG. All-poly tibial component better than metal-backed: a randomized RSA study. Knee. 2004 Jun;11(3):189-96. doi: 10.1016/S0968-0160(03)00071-1. PMID 15194094
- [Background] Nouta KA, Verra WC, Pijls BG, Schoones JW, Nelissen RG. All-polyethylene tibial components are equal to metal-backed components: systematic review and meta-regression. Clin Orthop Relat Res. 2012 Dec;470(12):3549-59. doi: 10.1007/s11999-012-2582-2. Epub 2012 Sep 13. PMID 22972656
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075